CLINICAL TRIAL: NCT03561454
Title: A Registry of Intra-Operative Radiation Therapy (IORT) Using the Xoft ® Axxent ® eBx™ System Patients
Brief Title: A Registry of Intra-Operative Radiation Therapy (IORT) Using the Xoft ® Axxent ® eBx ™ System Patients
Status: Active, not recruiting | Type: Observational
Sponsor: MedStar Franklin Square Medical Center (Other)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20180335
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-03

CONDITIONS: Early Stage Breast Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: IORT — Intra-Operative Radiation Therapy

SUMMARY:
Single arm, prospective, multi-center, non-randomized study of subjects treated with single fraction, intra-operative radiation therapy at the time of lumpectomy for early stage breast cancer.To assess the rate of ipsilateral breast tumor recurrence in subjects treated with the Xoft Axxent Electronic Brachytherapy System when used for single-fraction, intra-operative radiation therapy treatment of early stage breast cancer when compared to whole breast irradiation (WBI) at 5 years of follow-up. The results of this single arm study will be compared to whole breast irradiation (WBI).

ELIGIBILITY:
General Inclusion Criteria

1. Subject must have provided written Informed Consent
2. Subject must have biopsy-proven ductal carcinoma in situ (DCIS) or invasive ductal carcinoma of the breast

   a. In addition to invasive ductal carcinoma, allowable invasive carcinomas are: i. Adenoid cystic (or adenocystic) carcinoma ii. Low-grade adenosquamous carcinoma iii. Medullary carcinoma iv. Mucinous (or colloid) carcinoma v. Papillary carcinoma vi. Tubular carcinoma vii. Metaplastic carcinoma viii. Micropapillary carcinoma ix. Mixed carcinoma
3. Subject must be female ≥ 40 years of age
4. Subject's tumor(s) must be < 3.0 cm in greatest diameter by pre-operative assessment
5. Clinical staging of Subject's tumor(s) must meet AJCC Tumor Classification: Tis, T1 or T2 (< 3 cm), N0, M0
6. Subject presenting with bilateral breast cancer may be enrolled if BOTH cancers meet all of the inclusion and none of the exclusion criteria
7. Women of child-bearing potential must have a negative pregnancy test within one week of IORT treatment
8. Women of child-bearing potential must agree to use adequate contraceptive precautions (defined as intrauterine devices, surgical contraceptives or a combination of condom and spermicide) from the time of negative pregnancy test through completion of the radiation treatment period

General Exclusion Criteria

1. Subject is pregnant or nursing
2. Subject has significant auto-immune disease
3. Subject has a pacemaker present in the field of radiation or quadrant of the breast cancer
4. Subject has multi-focal breast cancer where the sum of the individual tumor sizes (greatest diameters) are > 3 cm Subject has multi-centric breast cancer
5. Subject has known lympho-vascular invasion
6. Subject has invasive lobular cancer
7. Subject has undergone neo-adjuvant chemotherapy or neo-adjuvant endocrine therapy for current breast cancer
8. Subject has a history of recurrent breast cancer in the ipsilateral breast
9. Subject has had previous radiation exposure of the involved breast
10. Subject has BRCA 1 or 2 mutations. Note: Testing will only be required for subjects presenting with bilateral breast cancer; testing is not required for unilateral cancers
11. Subject has contraindications for radiation
12. Subject considered by the Investigator to be high-risk for breast conservation surgery and/or intra-operative radiation therapy
13. Subject has participated in any other clinical investigation that is likely to confound study results or affect study outcome either at the time of IORT or for 3 months prior to IORT

Ages: 40 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female 40 years of age and older receiving IORT treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
tumor recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Maen Farha, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Good Samaritan Hospital, Baltimore, Maryland, United States